CLINICAL TRIAL: NCT04669418
Title: Host RNA Signature to Discriminate Bacterial From Viral Infection and Non-specific Inflammation in Children With Cancer
Brief Title: Host RNA Signature in Children With Cancer and Infection
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Børnecancerfonden (Other); Lundbeck Foundation (Other); Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Lotte Møller Smedegaard, M.D., Rigshospitalet, Denmark
Other Study IDs: H-2-2010-002_1
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Childhood Cancer; Infection; Neutropenia, Febrile
MeSH Terms: conditions — Neoplasms; Infections; Febrile Neutropenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All children will have 2.5 ml whole blood drawn into a PaxGene RNA (Qiagen®) tube along with routine blood tests. Only RNA is extracted
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: 70 children with cancer and a positive blood culture.
  Interventions: Diagnostic Test: RNA expression signature
- Group 2: 50 children with cancer and no positive blood culture.
  Interventions: Diagnostic Test: RNA expression signature

INTERVENTIONS:
Diagnostic Test: RNA expression signature — Whole transcriptome profiling using RNA sequencing

SUMMARY:
The aim is to investigate if RNA expression signature can discriminate bacterial from viral infection or non-infectious inflammation in children with cancer.

Earlier studies in immunocompetent children have shown promising results, but studies in immunocompromised children are lacking.

We aim to include 300 febrile episodes in children with cancer. The samples will be analysed by RNA sequencing. If succesfull, this method can help prevent unnecessary antibiotic treatment, reduce hospital admissions, side effects and antimicrobial resistance and improve quality of life for children during cancer treatment.

DETAILED DESCRIPTION:
Children with cancer are at high risk of invasive bacterial infections particularly during neutropenia. Febrile neutropenia is an early sign of a potentially fatal infection requiring broad-spectrum empiric antibiotics. However, the majority of children do not have a bacterial infection, but still receive antibiotics, since current tests cannot distinguish causes of fever. A number of transcriptomic studies of immunocompetent patients show that host leukocyte patterns of activated RNA can discriminate bacterial infection from non-infectious inflammation with high accuracy, but studies in immunocomprised patients are few.

Methods

A prospective non-interventional observational multicentre study including febrile childhood cancer patients during 24 months at all Danish Pediatric Oncology Departments (Rigshospitalet, Aarhus, Odense and Aalborg University Hospitals). Leukocyte RNA expression will be analysed in whole blood samples by RNA sequencing adjusted for low RNA input. 300 febrile episodes will be included, and predictive host RNA signatures will be identified in a discovery cohort and assessed in a validation cohort. Further, to explore the transcriptome in non-febrile children with neutropenia, we include a control group of 15 children with cancer and no fever.

Time frame Inclusion of children: 1st of June 2019 to 31st of May 2021 Analysis of samples (RNA sequencing): 1st of June 2021 - 1st of December 2021

Perspective

The study will create a base for a randomised trial regarding implementation of RNA signature versus normal procedure in handling febrile children with cancer. This can lead to the development of a targeted RNA-expression analytical platform that can prevent unnecessary antibiotic treatment in the majority of children with febrile neutropenia. This will reduce hospital admissions, side effects, antimicrobial resistance and improve quality of life during cancer treatment. The results can be extrapolated to the adult patients with cancer, who are often treated with prophylactic antibiotics, which complicate finding the infectious agent. Additionally, the test may be applied in other immunosuppressed children with infections.

ELIGIBILITY:
Inclusion Criteria:

Children with cancer and fever. Fever defined as temperature above 38.5 °C measured once, or 38.0-38.5 °C for ≥ 1 hour.

Exclusion Criteria:

The children can be excluded if they turn out to have a different diagnosis than expected or if it is not possible to draw the blood tests.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cancer and fever admitted to the Pediatric Oncology Departments throughout Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
RNA signature | 1.5 years
  To detect specific RNA signatures in whole blood in children with febrile neutropenia

SECONDARY OUTCOMES:
Time study | 1,5 years
  An investigation of the change in RNA expression over time during an infection period
Application of known RNA signatures | 1,5 years
  To test RNA signatures from genes published in other studies eg. the genes IFI44L and FAM89A
Differences in RNA signature according to pathogen | 1,5 years
  To investigate potential differences in RNA signatures in patients with gram positive versus gram negative bacteria
Comparishment of RNA signatures in neutropenic and non-neutropenic children | 1,5 years
  To compare RNA signatures in febrile neutropenic and non-neutropenic children with a positive blood culture

CONTACTS AND LOCATIONS:
Overall Officials: Lotte M. Smedegaard, M.D., Principal Investigator — ph.d.-student
Locations (5):
- Denmark (5):
  - Department of Pediatrics, Aalborg University Hospital, Aalborg
  - Department of Pediatric Oncology, Aarhus University Hospital, Aarhus
  - Center for Genomic Medicine, Copenhagen
  - Department of pediatric and adolescent medicine, Rigshospitalet (Copenhagen University Hospital), Copenhagen
  - Department of Pediatrics, The H.C. Andersen's Children's hospital, Odense

IPD SHARING:
Plan to Share IPD: Undecided